CLINICAL TRIAL: NCT02931318
Title: The Knowledge Levels and Attitudes of the People Living in the City Center of Nevşehir on Organ Donation and Transplantation
Brief Title: The Knowledge Levels and Attitudes of the People Living in Nevşehir on Organ Donation and Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nevsehir Public Hospital (Other Government)
Collaborators: Nevsehir Haci Bektas Veli University (Other)
Responsible Party: Principal Investigator, Mehmet Akif Yazar, Responsible of Critical Care, Nevsehir Public Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 02/01
Record Dates: First submitted 2016-05-28; First posted 2016-10-13 (Estimated); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Organ Finding
Keywords: Organ donation; brain death; public opinion
MeSH Terms: conditions — Brain Death

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nevsehir (Experimental): People Living in the City Center of Nevşehir
  Interventions: Behavioral: Nevsehir

INTERVENTIONS:
Behavioral: Nevsehir — The data of the study were collected with the questionnaire

SUMMARY:
In this descriptive study, the purpose was to determine the knowledge levels and attitudes of the people in Nevsehir, Turkey on organ donation.

It has been determined that the people living in Nevsehir do not have sufficient knowledge on organ donation, they had various concerns on the issue, and they wanted to receive information from Organ Donation Units. It can be used the exemplification and internalization in educational curricula about increasing the organ donation.

DETAILED DESCRIPTION:
Purpose

In this descriptive study,the purpose was to determine the knowledge levels and attitudes of the people in Nevsehir on organ donation.

Methods

The data of the study were collected with the questionnaire applied to 414 people residing in Nevşehir between February and May 2016. In evaluating the data, the numbers, percentage calculations, Chi-Square Test,t-test, and One-Way tests were used.

ELIGIBILITY:
Inclusion Criteria:

* Anyone aged between 20-65
* The people living in the city center of Nevşehir, Turkey

Exclusion Criteria:

* <20 years old

  * 65 years old
* The people who do not live the city center of Nevşehir, Turkey

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 414 (Actual)
Dates: Start 2016-02; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Questionnaire | 3 months
  the knowledge levels of the people in Nevsehir, Turkey on organ donation.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Akif Yazar, MD, Principal Investigator — republic of turkey ministry of health

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Haustein SV, Sellers MT. Factors associated with (un)willingness to be an organ donor: importance of public exposure and knowledge. Clin Transplant. 2004 Apr;18(2):193-200. doi: 10.1046/j.1399-0012.2003.00155.x. PMID 15016135
- [Result] Sanner MA. A Swedish survey of young people's views on organ donation and transplantation. Transpl Int. 2002 Dec;15(12):641-8. doi: 10.1007/s00147-002-0474-1. Epub 2002 Nov 5. PMID 12478412